CLINICAL TRIAL: NCT04627987
Title: Mechanisms of Excess Risk in Aortic STEnosis After Aortic Valve Replacement
Brief Title: Mechanisms of Excess Risk in Aortic Stenosis
Acronym: MASTER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 125312
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Aortic Stenosis; Non-Sustained VT; Heart Failure
Keywords: Late gadolinium enhancement; Tissue characterisation; Arrhythmia; Sudden cardiac death; Heart failure; Aortic stenosis; Myocardial remodelling
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure; Arrhythmias, Cardiac; Death, Sudden, Cardiac | interventions — Walk Test; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Myocardial biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main study: Patients with severe, symptomatic aortic stenosis will be recruited and followed up with primary outcome of heart failure death and hospitalisation (n=192). Of these, 170 will have an implantable cardiac monitor placed to detect presence and burden of non-sustained VT.
  Interventions: Diagnostic Test: Cardiac MRI scan; Diagnostic Test: Serum biomarkers (High sensitivity troponin, NT-proBNP; Procedure: Implantable Loop Recorder; Diagnostic Test: 6 minute walk test; Diagnostic Test: Echocardiogram

INTERVENTIONS:
Diagnostic Test: Cardiac MRI scan — Cardiac MRI scan pre- and post- aortic valve replacement to assess degree of left ventricular remodelling, fibrosis and myocardial blood flow.
Diagnostic Test: Serum biomarkers (High sensitivity troponin, NT-proBNP — Blood tests looking evidence of cardiac structural remodelling and function.
Procedure: Implantable Loop Recorder — Determine post-AVR arrhythmia burden
Diagnostic Test: 6 minute walk test — Validated assessment of functional capacity - distance walked over 6 minute time frame.
Diagnostic Test: Echocardiogram — Ultrasound assessment of heart structure and function. Standard of care in valve surgery pathway.

SUMMARY:
Aortic stenosis (AS) is caused by narrowing of one of the main heart valves. Replacing the valve is the only treatment to prevent the heart from failing or death. The timing of replacement is currently often too late - half of patients are left with permanent scarring and a quarter die within 3.5 years.

Studies are underway to see if earlier replacement makes a difference. But for those with scarring of the heart, there is currently no tailored treatment. I want to change this by understanding why and how patients with scar are dying and what the investigators can do to prevent this.

In this study, the investigators will use a heart scan (MRI) to detect scarring before valve replacement. After replacement, patients will receive a tiny monitor (paper clip size), which the investigators inject underneath the skin. This monitor continuously checks the heartbeat and can detect increased body fluid due to heart failure. The investigators will monitor patients for an average of 3 years to see if scarring is linked to abnormal heart rhythms and heart failure.

Once the investigators know how and why, the investigators can target patients with available medications and design studies using specialised treatments, eg defibrillator implantation, to protect patients with scar from dying.

DETAILED DESCRIPTION:
Valvular heart disease (VHD) affects around 1.5 million people above the age of 65 across the UK and is set to nearly double by 2050. Aortic Stenosis (AS) is the most common VHD in the UK, affecting 3% of those over 75 with more than 11,000 people requiring aortic valve replacement (AVR) in the UK each year (>100,000 world-wide). Current guidelines recommend AVR to improve survival and symptom status when AS symptoms emerge or there is a reduction in left ventricle (LV) function (1), but years of excessive haemodynamic load result in an "AS cardiomyopathy" with LV hypertrophy, remodelling, diffuse and focal scar. The investigators, and others, have shown that these changes lead to an excess in morbidity and mortality, but the mechanisms of increased risk is unclear.

Patients undergoing aortic valve replacement for severe aortic stenosis have a shorter life expectancy compared with the general population (2). Years of excessive haemodynamic load result in an "AS cardiomyopathy" with LV hypertrophy, remodelling, diffuse and focal scar. The investigators and others have shown that these changes to the heart muscle are associated with poor outcome. But the mechanism of how heart muscle damage leads to excess mortality is poorly understood.

The proposed study will enhance our understanding of the residual risk after AVR and reveal the modes and substrate of mortality. Heart failure and heart rhythm disturbances (arrhythmias) are likely downstream effects of heart muscle damage, but without understanding the mode of death (heart failure, arrhythmia or other), the investigators are unable to target therapeutic strategies to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic severe aortic stenosis referred for surgical or transcatheter AVR (one out of: effective orifice area [EOA] <1.0 cm2 , indexed EOA of 0.6cm/m2, peak velocity >4.0 m/s or mean gradient >40mmHg).

Exclusion Criteria:

* More than moderate valve disease other than AS
* Diagnosis of dilated or hypertrophic cardiomyopathy, pregnancy/breast feeding
* eGFR <30ml/min, CMR incompatible devices
* Inability to complete the protocol
* Other conditions that would prevent participation in the study.
* Adenosine perfusion will not be performed in patients with AV block, severe asthma/COPD or LVEF<40%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective single centre, observational cohort study of patients with symptomatic severe AS (n=192) undergoing clinically indicated AVR (surgical or transcatheter) and multiparametric assessment by CMR prior to AVR.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Heart failure death or hospitalisation for heart failure. | 5 years after aortic valve replacement
Burden of non-sustained VT | 2.5 years after aortic valve replacement.
  As assessed on implantable cardiac monitor (approximate battery life 2.5 years)

SECONDARY OUTCOMES:
All-cause mortality (all-cause and cardiovascular via NHS spine/death registration) | 5 years after aortic valve replacement
change in functional capacity (6-minute walk test) | At 6 weeks and 12 months after aortic valve replacement.
Heart failure symptoms | At 6 weeks and 12 months post aortic valve surgery
  New York Heart Association (NYHA) functional classification (NYHA 1 least symptomatic, 4 most symptomatic)
Heart failure symptoms | At 6 weeks and 12 months post aortic valve surgery
  World Health Organisation Disability Assessment Schedule 2.0 (Higher score indicates greater disability)
Burden of other serious arrhythmias requiring change in management | 2.5 years after aortic valve replacement
  Participants with complete heart block, Mobitz 2 AV block, new onset atrial fibrillation

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bennett J, Thornton GD, Nitsche C, Gama FF, Aziminia N, Gul U, Shetye A, Kellman P, Davies RH, Moon JC, Treibel TA; Barts Valve and Imaging Group. Left Ventricular Hypertrophy in Aortic Stenosis: Early Cell and Matrix Regression 2 Months Post-Aortic Valve Replacement. Circ Cardiovasc Imaging. 2024 Dec;17(12):e017425. doi: 10.1161/CIRCIMAGING.124.017425. Epub 2024 Dec 4. PMID 39629586